CLINICAL TRIAL: NCT02338570
Title: Outcome-related Factors in Patients With Metastatic Renal Cell Carcinoma Treated With Everolimus After Failure of a First-line Treatment With VEGF Inhibitor
Brief Title: Outcome-related Factors in Patients With Metastatic Renal Cell Carcinoma Treated With Everolimus (ORCHIDEE)
Acronym: ORCHIDEE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped on November 16th 2016, because of recruitment failure.
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRFMN-RCC-6691
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2016-11

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Other): All patients will receive everolimus 10 mg orally per day. Treatment will continue until progression, unacceptable toxicity, patient refusal or medical decision
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Patients will start study treatment on day 1 and will be treated with daily doses of everolimus (10 mg daily tablets).
  Other Names: Afinitor

SUMMARY:
Evaluation of unfavourable outcome-related factors in patients affected by renal cell cancer in treatment with everolimus and previously treated with a Vascular endothelial growth factor (VEGF) inhibitor (i.e. sunitinib, sorafenib,pazopanib, or bevacizumab+interferon)

DETAILED DESCRIPTION:
Predictive factors to be considered are: histology, Heng risk group, Eastern Cooperative Oncology Group-performance status (ECOG-PS), site of metastases, glycemia and cholesterolemia.

The data collected in this "real life" population could contribute to identify clinical factors that predict favourable outcomes in patients treated with everolimus after failure or a a first-line treatment with a VEGF inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years or older, with histologically or cytologically confirmed mRCC (clear cell or not clear cell);
2. ECOG-PS 0-1-2;
3. With target and/or non-target lesions according to Response Evaluation Criteria In Solid Tumours (RECIST) 1.1;
4. Following failure of a previous treatment with VEGF-targeted therapy (e.g. sunitinib, sorafenib, pazopanib, or bevacizumab+interferon);
5. For whom a decision has been taken to initiate everolimus treatment or patient currently receiving treatment with everolimus by a period of time ≤30 days;
6. Willing and able to comply with follow-up and all other protocol requirements and able to commence treatment within 21 days;
7. Written informed consent obtained before any screening procedure and according to local guidelines.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Previous treatment with everolimus or at the date of written informed consent provision receiving everolimus by more than 30 days;
2. Symptomatic central nervous system metastases. Patients may be eligible if the central nervous system metastases have been adequately treated (surgery or radiotherapy), and do not require ongoing corticosteroids for control of symptoms and have had no evidence of progression for at least three months;
3. Other malignancy diagnosed within the last 5 years, except the following, if adequately treated: superficial squamous cell carcinoma or basal cell carcinoma of skin, superficial bladder cancer (T1 and G1 or T1 and G2), stage 1 cervical cancer;
4. Treatment with an investigational agent in the past 4 weeks;
5. Clinically relevant human immunodeficiency virus, hepatitis B virus, hepatitis C virus infection;
6. Non adequate liver function as shown by:

   * serum or plasma ALT and AST >3.0x upper limit of normal (ULN) >5 if hepatic metastases are present;
   * Serum or plasma total bilirubin: >1.5xULN (excepted for patients with Gilbert's syndrome);
7. Non adequate renal function as shown by serum creatinine >2.5xULN;
8. Any of the following in the last year: myocardial infarction, severe/ unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack or pulmonary embolism;
9. Ongoing grade ≥2 cardiac dysrhythmias, atrial fibrillation of any grade or prolongation of the corrected QT interval to >450 msec for males or >470 msec for females;
10. Pregnancy (negative pregnancy test required for women of child-bearing potential), breast feeding;
11. Inadequate contraception. Women must be post-menopausal, surgically sterile, or use a reliable form of contraception. Men must be surgically sterile or use a barrier method of contraception;
12. Known allergy or hypersensitivity to everolimus or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
predictive factors identification | 36 months
  To identify factors predictive of a favourable outcome, in terms of survival free from an unfavourable event, in patients treated with everolimus as second line treatment for metastatic renal cell carcinoma (mRCC). A favourable outcome is being alive and on treatment without both disease progression (according to RECIST 1.1) and HRQoL deterioration (7-point decrease from baseline evaluation on the EQ-5D VAS).

SECONDARY OUTCOMES:
Progression free survival (PFS) of everolimus as second line treatment | 36 months
  PFS distributions will be estimated using the Kaplan-Meier method and compared using the log-rank test.
health related quality of life (HRQoL) | 36 months
  As measured by EQ-5D questionnaire. It will be described at each time by using summary statistical measures for continuous variables
drug-related toxicity | 36 months
  assessed by the National Cancer Institute-Common Terminology Criteria for adverse events (NCI-CTCAE), version 4.03.
  The frequency of maximum toxicity grade experienced by each patient for each specific toxicity will be presented as well as the frequency of patients experiencing grade 3 or 4 (grade 2 for neurotoxicity) events, and SADRs.
compliance | 36 months
  Treatment compliance will be assessed by evaluating the dose intensity (total dose divided by duration of exposure to treatment in weeks), and calculating the frequencies and proportion of patients who modified or interrupted the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Cartenì, Principal Investigator — Azienda Ospedaliera "Antonio Cardarelli", Napoli
Locations (8):
- Italy (8):
  - Spedali Civili, Brescia
  - Ospedale A Perrino, Brindisi
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale, Napoli
  - AOU Maggiore della Carità, Novara
  - Casa di Cura La Maddalena, Palermo
  - Unicampus Biomedico, Roma
  - AOU San Giovanni di Dio e Ruggi D'Aragona, Salerno